CLINICAL TRIAL: NCT04019392
Title: The Rate of Intramuscular Tissue Temperature Reduction Between Wetted Ice With Elastic Wrap and Game Ready
Brief Title: Rate of Tissue Temperature Reduction Between Wetted Ice and Game Ready
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Dakota State University (Other)
Responsible Party: Principal Investigator, Kara Gange, Associate Professor, North Dakota State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HE20001
Record Dates: First submitted 2019-07-10; First posted 2019-07-15 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Cryotherapy Effect
Keywords: cooling rates

STUDY DESIGN:
Intervention Model Description: A 2 x 4 repeated measures design to determine decreases in triceps surae intramuscular tissue temperature will be used for this study. The independent variables will be the cryotherapy modalities (Game Ready® and wetted ice bag with elastic wrap) and time (baseline, 10 minutes, 20 minutes, and 30 minutes). The dependent variable will be the medial triceps surae intramuscular tissue temperature.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Wetted ice with elastic wrap (Active Comparator): A standard ice bag filled with 2000 mL of cubed ice and 300 mL of 5˚C water will be applied to each participants' lower leg for 30 minutes using an elastic wrap. The elastic wrap will be applied at approximately 75% percent tension starting distal to the treatment area and moving proximally overlapping by half. The elastic wrap application will consist of pulling the wrap to its full tension, measuring the length of the wrap, and calculating 75% of the total length to apply to the body part.
  Interventions: Device: Game Ready® device
- Game Ready (Active Comparator): The half leg boot sleeve of the Game Ready® device (CoolSystems, Inc., Alamda, CA) will be applied to each participants' lower leg and ankle for 30 minutes set on the medium pressure setting (5-50 mmHG).
  Interventions: Other: Wetted Ice Bag with Elastic Wrap

INTERVENTIONS:
Device: Game Ready® device — The half leg boot sleeve of the Game Ready® device (CoolSystems, Inc., Alamda, CA) will be applied to each participants' lower leg and ankle for 30 minutes set on the medium pressure setting (5-50 mmHG).
  Arms: Wetted ice with elastic wrap
Other: Wetted Ice Bag with Elastic Wrap — A standard ice bag filled with 2000 mL of cubed ice and 300 mL of 5˚C water will be applied using an elastic wrap to each participants' lower leg for 30 minutes. An elastic wrap applied at approximately 75% percent tension starting distal to the treatment area and moving proximally overlapping by half will be applied over the wetted ice bag.
  Arms: Game Ready

SUMMARY:
This study compares the tissue temperature decrease between a wetted ice bag (ice and water) with an elastic wrap to the Game Ready® treatment. The goal is to determine which one decreases the temperature the most and the fastest, which is important in immediate care treatments of a musculoskeletal injury.

DETAILED DESCRIPTION:
The purpose of this study will be to determine which cryotherapy method, wetted ice bag and elastic wrap or Game Ready® set at medium pressure, decreases tissue temperature the most during a 30-minute treatment. Due to the convenience of Game Ready®, it is being used as an immediate care intervention. Findings in the literature have indicated wetted ice cools tissue temperature more than cubed or crushed ice based on the assumption that colder is better. Conversely, research on Game Ready® has revealed ice bags and slush buckets cause a greater reduction in tissue temperature compared to Game Ready®. However, no study exists comparing the effects of Game Ready® versus wetted ice on intramuscular tissue temperature reduction as immediate care interventions. Based on the results, this study may help contribute to the existing literature on tissue temperature reduction of both Game Ready® and wetted ice to determine the better modality to use for immediate care. The research questions guiding this study will be:

1. Which cryotherapy method, Game Ready® or wetted ice with elastic wrap, will be the most effective at decreasing intramuscular tissue temperature during a 30-minute application in patients aged 18-40 years old?
2. Which cryotherapy method, Game Ready® or wetted ice with elastic wrap, will achieve an intramuscular tissue temperature reduction the fastest?

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be both male and female.
* Subjects will be between 18 and 40 years of age.
* Subjects will have no prior injury to the dominant lower leg within the past 6 months.
* Subjects will be able to speak English.
* Subjects will have less than 1 cm of adipose over the medial gastrocnemius muscle.

Exclusion Criteria:

* any current lower extremity injury, or any lower extremity injuries within the past 6 months.
* any previous history of surgery in the lower leg
* any contraindications to cryotherapy such as Raynaud's phenomenon, cold-induced urticaria, previous frostbite to the lower leg, open wounds, peripheral vascular disease, lupus, circulatory insufficiency, mayocardial ischemia, or skin infections.
* any abnormalities seen in the muscle as determined by diagnostic ultrasound.
* any allergies or sensitivities to Betadine.
* greater than 1.0cm of adipose over the medial gastrocnemius muscle (calf).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Intramuscular temperature | The tissue temperatures will be recorded every 5 seconds and analyzed at the baseline.
  The triceps surae intramuscular tissue temperature will be recorded with thermocouples inserted 2cm below the adipose.
Intramuscular temperature | The tissue temperatures will be recorded every 5 seconds and analyzed at 10 minutes.
  The triceps surae intramuscular tissue temperature will be recorded with thermocouples inserted 2cm below the adipose.
Intramuscular temperature | The tissue temperatures will be recorded every 5 seconds and analyzed at 20 minutes.
  The triceps surae intramuscular tissue temperature will be recorded with thermocouples inserted 2cm below the adipose.
Intramuscular temperature | The tissue temperatures will be recorded every 5 seconds and analyzed at 30 minutes/end time.
  The triceps surae intramuscular tissue temperature will be recorded with thermocouples inserted 2cm below the adipose.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Gange, PhD, ATC, Principal Investigator — Kara Gange
Locations (1):
- North Dakota State University, Fargo, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No